CLINICAL TRIAL: NCT07162142
Title: Retrograde Elastic Nailing With Pollar K-wire in Metaphyseal Diaphyseal Fracture of Distal Radius in Pediatric Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, abdalaziz youssef mohammed abdalhady, Principal Investigator, Al-Azhar University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RENPKMDFDRP
Record Dates: First submitted 2025-02-08; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Distal Radius Fracture
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- metaphyseal diaphyseal fracture of distal radial fracture in pediatrics (Experimental)
  Interventions: Procedure: elastic nailing with pollar K.wire

INTERVENTIONS:
Procedure: elastic nailing with pollar K.wire — retrograde elastic nailing of metaphyseal diaphyseal fracture of distal radius in pediatrics

SUMMARY:
Distal radius fractures are the most common fractures in the pediatric population . It accounts for 35% of all pediatric fractures . Although pediatric distal radius fractures can be successfully treated conservatively, reduction losses of 21-39% can be observed in the treatment with a plaster cast . Reduction losses are frequently observed in distal radius diaphyseal metaphyseal junctional (DRDMJ) fractures, primarily due to the limited contact surface of the fracture . There has yet to be a consensus regarding the treatment protocol for DRDMJ fractures . In DRDMJ fractures, surgery is recommended in cases where satisfactory alignment cannot be achieved with closed re-duction and cast immobilization, or there is reduction loss in clinical follow-ups .

ELIGIBILITY:
Inclusion Criteria:

- all distal radial fractures in pediatric patients 3-15 years failed closed reduction

Exclusion Criteria:

* pathological fracture

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0, Change From Baseline in Pain Scores on the Visual Analog Scale at 6 Weeks | three months

CONTACTS AND LOCATIONS:
Locations (1):
- Abdalaziz Youssef Mohammed, Cairo, Egypt